CLINICAL TRIAL: NCT01591564
Title: Interpersonal Psychotherapy in Youth With Severe Mood Dysregulation-Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Leslie Miller, M.D., Assistant Professor, Johns Hopkins University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00046454; K23MH090246 (NIH)
Record Dates: First submitted 2012-05-02; First posted 2012-05-04 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Severe Mood Dysregulation
Keywords: interpersonal psychotherapy; severe mood dysregulation
MeSH Terms: interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- therapy (Other): All participants will receive the intervention.
  Interventions: Behavioral: Interpersonal Psychotherapy for youth with SMD (IPT-SMD)

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy for youth with SMD (IPT-SMD) — Youth will receive weekly therapy sessions for 16 weeks and then bi-weekly session until week 20. Parent sessions will also be included.

SUMMARY:
The purpose of this study is to determine the feasibility and acceptability of an utilizing an adapted form (IPT-SMD)of a psychosocial intervention, Interpersonal Psychotherapy for Depressed Adolescents, for youth with severe mood dysregulation (SMD).

The investigators hypothesize that retention rates will be >80%,satisfaction scores will average 6 (high) on a 7 point satisfaction scale, and that youth who receive the IPT-SMD intervention will have overall improvement in SMD symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, ages 13 to 17 years, who meet criteria for severe mood dysregulation as defined by NIMH criteria.
* Subject has an estimated IQ >70 on the Kaufman Brief Intelligence Test (KBIT-2)
* Subjects will have continuously resided with a legal guardian who has known the adolescent well for at least one year before study entry and is legally able to sign the consent form.
* Participants must be on the same dose of any prescribed medication for 4 weeks prior to randomization.
* Children's Global Assessment Scale (CGAS) ≤ 60

Exclusion Criteria:

* Subject poses a significant risk for dangerousness to self or others. Risk will be determined by clinical history, clinical diagnostic interview and KSADS-PL interview of parent and patient by clinician.
* Subject suffers from a concomitant medical or psychiatric co-morbidity that makes this study protocol inadvisable (either the treatment is contraindicated or the disorder is not the primary focus of treatment).
* Subject meets DSM-IV criteria for current alcohol or substance dependence or current use (defined as the past 4 weeks).
* Pregnant females.
* Primary caretaker does not speak English

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2012-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Retention rate | 20 weeks
  We are assessing the feasibility and acceptability of IPT-SMD in anticipation of conducting a larger trial.

SECONDARY OUTCOMES:
Clinical Global Impressions Scale CGI-I (SMD) | 20 weeks
  We will utilize the CGI-I (SMD) to assess the effectiveness of IPT-SMD on the severity of SMD symptoms in youth with SMD.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Miller, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States